CLINICAL TRIAL: NCT01480947
Title: The Treatment Effect of Bio-Three on Children With Enteritis Due to Salmonella or Rotavirus or Any Unknown Reason
Brief Title: The Treatment Effect of Bio-Three on Children With Enteritis
Acronym: Bio-three
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yung-Feng Huang, Consultant Physician, Department of Pediatrics, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS98-CT1-11
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Gastroenteritis; Diarrhea
Keywords: probiotics; pediatric; salmonella; rotavirus; gastroenteritis
MeSH Terms: conditions — Gastroenteritis; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bio-Three (Experimental): add-on treatment of the probiotics (Bio-three)
  Interventions: Drug: Bio-three
- control treatment (No Intervention): control treatment (intravenous fluid, oral rice and half strength milk formula)
  Interventions: Drug: Bio-three

INTERVENTIONS:
Drug: Bio-three — oral Bio-three three times daily for 7 days, Bio-three dosage plan: 1) patients aged 6 years old, 1 tablet t.i.d.; 2) patients aged between 6 and 12 years old, 2 tablets t.i.d.; 3) patients aged 12 years old, 3 tablets t.i.d.

SUMMARY:
Diarrhea due to acute enteritis is a common symptom in the children. Lots of patients are infected by rotavirus or salmonella.

Base on the past researches, there is benefit effect of probiotics on patients with diarrhea or acute enteritis. In this clinical study, bio-Three, a probiotic which contains three independent probiotics, will be used in patients with acute diarrhea.

This is a single site, controlled clinical research. About 80 patients will be enrolled into this study to evaluate the benefit effect of bio-Three among patients with acute enteritis due to rotavirus or salmonella or other unknown reason. Patients will be diagnosed and screened by inclusion and exclusion criteria and only eligible patients will be enrolled into this study.

DETAILED DESCRIPTION:
Intervention: Subjects were randomly assigned to receive control treatment (intravenous fluid, oral rice and half strength milk formula) or add-on treatment of the probiotics (Bio-three®) to the control treatment.

Main outcome measures: Quantitative Vesikari scales and qualitative severe diarrhea (Vesikari scale≥11) Exclusion criteria included immunodeficiency, severe abdominal distension with risk of bowel perforation, severe infection or sepsis, history of gastrointestinal tract surgery, and probiotics use in the preceding 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptom of diarrhea less than 3 days

Exclusion Criteria:

* Severe abdominal distension with risk of bowel perforation
* Risk for sepsis
* Past history with surgical operation of gastrointestinal tracts
* immunodeficiency
* probiotics use in the preceding 1 week

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Quantitative Vesikari scales and qualitative severe diarrhea | 7 days
  Quantitative Vesikari scales and qualitative severe diarrhea (Vesikari scale≥11) Severity of diarrhea was evaluated according to the following features: volume of stools, fecal consistency, and frequency. Other clinical symptoms or signs, including fever, vomiting, daily intake, dehydration, and treatment were also assessed

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Feng Huang, MD. MSc, Principal Investigator — Department of Pediatrics, Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan.
Locations (1):
- Department of Pediatrics, Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan